CLINICAL TRIAL: NCT04137588
Title: A Prospective of Efficacy and Safety of Use of Platinum Based Doublet Chemotherapy Plus Antiangiogenesis and Immune Checkpoint Inhibitors in Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of Use of Platinum Based Doublet Chemotherapy Plus Antiangiogenesis and Immune Checkpoint Inhibitors in Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jian Fang, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: 20191023
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Advanced Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Angiogenesis Inhibitors; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: antiangiogenesis 7.5mg/Kg q3w+pemetrexed 500mg/m2 q3w+ platinum 75mg/m2 q3w
  Interventions: Drug: Antiangiogenesis Agents
- Group B: immune checkpoint inhibitors 200mg q3w+pemetrexed 500mg/m2 q3w+platinum 75mg/m2 q3w
  Interventions: Drug: Immune checkpoint inhibitor
- Group C: antiangiogenesis 7.5mg/Kg q3w+immune checkpoint inhibitors 200mg q3w+pemetrexed 500mg/m2 q3w+platinum 75mg/m2 q3w
  Interventions: Drug: Antiangiogenesis Agents; Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Antiangiogenesis Agents — antiangiogenesis agents plus chemotherapy as first line treatment
  Groups: Group A; Group C
Drug: Immune checkpoint inhibitor — immune checkpoint inhibitor plus chemotherapy as first line treatment
  Groups: Group B; Group C

SUMMARY:
The purpose of this study is to explore the efficacy and safety of Use of Platinum Based Doublet Chemotherapy Plus Antiangiogenesis and Immune Checkpoint Inhibitors in Patients With Advanced Non-squamous Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent;
2. Non-squamous non-small cell lung cancer, newly diagnosed or previously not treated with systemic chemotherapy and / or epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors treatment;
3. Aged 18-75 years;
4. Eastern Cooperative Oncology Group (ECOG) score ≤ 2;
5. Survival is expected to exceed 12 weeks ;
6. Patients had a wild-type genotype (WT population; patients with EGFR or ALK genetic alterations were excluded)

Exclusion Criteria:

If any of the following criteria is met, the subject shall be excluded:

1. Squamous cell carcinoma (including adenosquamous carcinoma) and small cell lung cancer (including small cell carcinoma and non-small cell mixed lung cancer);
2. In the past 2 weeks, there have been systematic anti-tumor treatment including chemotherapy (including thoracic chemotherapy), radiotherapy (excluding radiotherapy of metastatic lesions outside the thoracic radiation field), targeted therapy, immunotherapy and biotherapy;
3. The subject had received anti-vascular endothelial growth factor (VEGF) small molecule tyrosine kinase inhibitors or monoclonal antibodies in the past 4 weeks;
4. Laboratory results:

   * White blood cell count <3 × 109 / L, neutrophil count <1.5 × 109 / L, platelet <75 × 109 / L, or hemoglobin <8g / dL;
   * Coagulation abnormalities (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time (APTT) > 1.5 ULN), with bleeding tendency or being treated with thrombolysis or anticoagulation;
   * Serum total bilirubin ≥1.5 ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 ULN in the absence of liver metastases; ALT or AST ≥5 ULN in liver metastases;
   * Serum albumin <30g / L;
   * Serum creatinine ≥ 1.5 ULN or creatinine clearance <40ml / min; • Urine routine urinary protein ≥ ++, or 24 hours urine protein ≥ 1.0 g;
5. Heart disease with significant clinical symptoms, such as: congestive heart failure, coronary heart disease with symptom, arrhythmia hardly be controlled by drugs, myocardial infarction in 6 months, or heart failure;
6. Imaging (CT or MRI) showed a tumor lesion 5 mm away from the large vessels, or the presence of invasive central vasculature of the central tumor; imaging (CT or MRI) showed significant cavitation or necrosis of the lung tumor; Other diseases that may cause haemoptysis;
7. Imaging (CT or chest radiograph) showed significant pneumothorax, fluid pneumothorax;
8. Obvious cough blood in 6 months, or daily hemoptysis amounted to half a teaspoon (2.5ml) or more;
9. Significant bleeding symptoms or with definite bleeding tendency within 12 months before randomization, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, occult blood ++ and above, intracerebral hemorrhage, vasculitis, or with congenital or acquired coagulopathy disorders;
10. Thrombosis, cancer thrombosis (including arteriovenous thrombosis, tumor thrombus, pulmonary embolism, transient ischemic attack, etc.) occurred within 12 months;
11. There are gastrointestinal obstruction, peptic ulcer, Crohn's disease, ulcerative colitis and other gastrointestinal diseases or other diseases may cause gastrointestinal bleeding or perforation;
12. Severe respiratory diseases, or need long-term oxygen, corticosteroid treatment of diseases such as chronic obstructive pulmonary disease, interstitial lung disease and respiratory failure;
13. Patients with uncontrolled central nervous system metastasis;
14. There are serious uncontrolled systemic diseases, such as nephrotic syndrome, infection, poorly controlled diabetes;
15. Patients with active HIV（human immunodeficiency virus）, HBV（hepatitis B virus）, or HCV（hepatitis C virus） infection;
16. Patients had undergone surgery (<28 days) or did not heal completely, or had other unhealed wounds before the study;
17. Patients known to be allergic to bevacizumab or any of the components of the drug;
18. Pregnant or lactating female patients, or unwilling to take contraceptive measures of reproductive age patients (including men);
19. There is a serious psychological or mental abnormality, or lack of compliance;
20. The investigator determines other circumstances that may affect the conduct of clinical studies and the determination of findings;
21. Participants with an active, known or suspected autoimmune disease;
22. Participants with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of first treatment;
23. Participants with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug related pulmonary toxicity.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Males and females, 18-75 years of age, non squamous non-small cell lung cancer, wild type genotype
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2021-03-03 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | one year
  ORR of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jian Fang, Beijing, Beijing Municipality, China